CLINICAL TRIAL: NCT03897582
Title: Beta-Lactams Dosing In Pneumonia in ICU in Patients Treated by Continuous Renal Replacement Therapy
Brief Title: Beta-Lactams Dosing In Pneumonia in ICU in Patients Treated by Continuous Renal Replacement Therapy: the BLIPIC Study
Acronym: BLIPIC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Valenciennes (Network)
Collaborators: Centre Hospitalier de Lens (Other); Centre Hospitalier de Bethune (Network); University Hospital, Lille (Other); General Hospital of Douai (Other); Centre hospitalier de Boulogne (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-05
Record Dates: First submitted 2019-03-07; First posted 2019-04-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Beta-lactam; Continuous Renal Replacement Therapy; Pneumonia; Antibiotic
Keywords: amoxicillin; amoxicillin-clavulanic acid; piperacillin-tazobactam; cefotaxime; ceftazidime; cefepime; meropenem; imipenem; multifiltrate; citrate; CVVHD; extended and continuous infusion; TDM; Therapeutic Drug Monitoring
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumonia are the most frequent infections in ICU. Little is known about beta-lactam doses necessary for this infection for patients treated with continuous veino-veinous hemodialysis. The pharmacokinetic variability expose to over and underdosage leading to toxicity or therapeutic failure. The aim of this study is to define if beta-lactams doses used in pneumonia for patients with acute kidney injury treated with our hemodialysis conditions lead to beta-lactam therapeutic plasma levels.

DETAILED DESCRIPTION:
Pneumonia are the most frequent infections in ICU. Little is known about beta-lactam doses necessary for this infection for patients treated with continuous veino-veinous hemodialysis. The pharmacokinetic variability expose to over and underdosage leading to toxicity or therapeutic failure. The aim of this study is to define if beta-lactams doses used in pneumonia for patients with acute kidney injury treated with our hemodialysis conditions lead to beta-lactam therapeutic plasma levels.

This prospective observational multicenter study will include all patients with pneumonia treated by beta-lactam and continuous veino-veinous hemodialysis in 5 ICU. Blood sampling will be done at assumed pharmacokinetic steady state. Protocol sample concentrations of beta-lactams immediately prior to re-dosing, after 24 hours of association of intraveinous beta-lactam and continuous veino-veinous hemodialysis. Another sample will be done after 48 hours. The ICU measured bacterial MICs routinely when the pathogen will be determined. Surveyed ICUs will adopt SFM-EUCAST breakpoints for the targeted (or suspected) bacteria to determine pharmacokinetic/pharmacodynamic targets when a mesured MIC (Minimum inhibitory concentration) is not available. Local hospital antibiogram data can also be used to describe likely pathogen susceptibility. Target attainment is defined as 100% fT> 5 MIC. Due to the long delay to receive therapeutic drug monitoring results, doses could not be ajusted. Factors which could cause concentrations variations will be registered. When neurotoxicity is suspected, a sample will be realized to know beta-lactam concentration and the adverse event will be notified.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Receiving intraveinous beta-lactam : amoxicillin, amoxicillin-clavulanic acid, piperacillin-tazobactam, cefotaxime, ceftazidime, cefepime, meropenem, imipenem
* With AKI defined as any of the following, and treated with Multifiltrate Ci-Ca CVVHD 1000® kit with a dialysis dose of 25 ml/kg/h :

  * Increase in creatininemia ≥ 0.3 mg/dl (≥ 26.5 µmol/l) within 48 hours
  * Increase in creatininemia ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days
  * Urine volume < 0.5 ml/kg/h for 6 hours
* Hospitalized in ICU
* Presence of a catheter to facilitate sample collection
* With pneumonia defined as any of the following :

  * Chest X-ray pneumonia : opacities, new or progressive infiltrates
  * AND at least one of the following : hyperthermia > 38°C or hypothermia < 36°C with no other explanation ; leukopenia < 4 G/L ou leukocytosis > 12G/L
  * AND at least one of the following : new onset purulent sputum or change in sputum character, new onset or worsening cough or dyspnea or tachypnea, rales or bronchial breathing, lower oxygen saturation/hypoxemia or increase of oxygen needs or respiratory assistance
* Treated within 24 hours by citrate hemodialysis AND beta-lactam respecting dose and administration conditions of the study :

  * Amoxicillin : loading dose followed immediately by 2g by extended infusion for 4 hours every 8 hours
  * Amoxicillin-clavulanic acid : 2g every 8 hours by intermittent bolus
  * Piperacillin-tazobactam: loading dose followed immediately by 4g/0.5g by continuous infusion every 8 hours (< 80 kg) ou 6 hours (> 80 kg)
  * Cefotaxime: loading dose followed immediately by 2g by continuous infusion every 8 hours Ceftazidime : loading dose followed immediately by 2g by continuous infusion every 8 hours
  * Cefepime: loading dose followed immediately by 2g by continuous infusion every 8 hours
  * Meropenem : loading dose followed immediately by 2g (> 60 kg) ou 1,33g (< 60 kg) by extended infusion for 4 hours every 8 hours
  * Imipenem : loading dose followed immediately by 750 mg (< 80 kg) ou 1g (> 80 kg) by extended infusion for 4 hours every 6 hours In case of extrem weight, dose will be on investigator's discretion but administration conditions have be to respected.
* No objection has been obtained from the patient or their legally authorised representative

Exclusion Criteria:

* Aged < 18 years
* ECMO
* Cystic fibrosis
* Burn victim
* Pregnant woman
* Any rapidly-progressing disease or immediately life-threatening illness
* Objection from the patients or their legally authorised representative
* No social security scheme
* Interruption of antibiotic before samples
* Patient in prison

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with pneumonia in ICU treated with intraveinous beta-lactams and CVVHD
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of beta-lactams concentrations above plasma therapeutic levels | Day 3 after start of antibiotic and continuous veino-veinous hemodialysis
  We aimed to obtain concentrations over 5 MIC (Minimum inhibitory concentration) for at least 80% of patients.

SECONDARY OUTCOMES:
Distribution of steady state beta-lactam concentrations and their variability | Day 3 after start of antibiotic and continuous veino-veinous hemodialysis
  Description of beta-lactam concentration
Incidence of neurotoxicity | Day 7 after start of antibiotic and continuous veino-veinous hemodialysis
  Percentage of neurotoxicity
Trends in beta-lactam concentrations between 2 days | At Day 1 and Day 2
  Comparaison between 24 hours and 48 hours samples
Clinical response observed when beta-lactam concentrations achieved 5 MIC | At Day 28 and day 90
  Survival at Day 28 and Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Lambiotte, MD, Study Chair — Centre Hospitalier de Valenciennes
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, Nord, France

REFERENCES:
- See also: SFAR, SFPT, Recommandations de Pratiques Professionnelles, Optimisation du traitement par bêta-lactamines chez le patient de soins critiques 2018. — https://sfar.org/optimisation-du-traitement-par-beta-lactamines-chez-le-patient-de-soins-critiques/